CLINICAL TRIAL: NCT03177681
Title: The Effect of Yogurt in Cancer Patient With Moderate Gastrointestinal (GI) Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 0 patient accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0052; NCI-2018-01356 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Malignant neoplasms of independent (primary) multiple sites; Gastrointestinal symptoms; Probiotics; Yogurt; Stool sample; Questionnaires; Surveys; Holter monitor
MeSH Terms: interventions — Medicine, Chinese Traditional; Surveys and Questionnaires; Electrocardiography, Ambulatory; Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Antibiotics Taken During Past 2 Weeks (Experimental): Group 1: Participant was on antibiotics anytime during the past 2 weeks prior to the time of enrollment.
  Tongue assessment, stool sample, and questionnaires done at baseline and once during Days 3-7 and once during Days 8-12.
  Participants wear a Holter monitor for 20-24 hours at baseline and once during Days 3-7 and once during Days 8-12.
  Participants given 2 tablespoons (33 cc) of yogurt each day for 12 days.
  Interventions: Other: Tongue Assessment; Other: Stool Sample; Behavioral: Questionnaires; Device: Holter Monitor; Other: Yogurt
- Group 2 - No Antibiotics Taken During Past 2 Weeks (Experimental): Group 2: Participant has not been on antibiotics in the past 2 weeks.
  Tongue assessment, stool sample, and questionnaires done at baseline and once during Days 3-7 and once during Days 8-12.
  Participants wear a Holter monitor for 20-24 hours at baseline and once during Days 3-7 and once during Days 8-12.
  Participants given 2 tablespoons (33 cc) of yogurt each day for 12 days.
  Interventions: Other: Tongue Assessment; Other: Stool Sample; Behavioral: Questionnaires; Device: Holter Monitor; Other: Yogurt

INTERVENTIONS:
Other: Tongue Assessment — The coating on the top of the tongue assessed and categorized into three categories: no coating, thin coating and thick coating. The coating of the tongue may be related to the microorganisms in the intestine.
Other: Stool Sample — Stool sample collected at baseline and once during Days 3-7 and once during Days 8-12.
Behavioral: Questionnaires — Participants complete 4 questionnaires about symptoms in the past 24 hours, irritable bowel syndrome (IBS), most recent stool, and quality-of-life. Questionnaires completed at baseline and once during Days 3-7 and once during Days 8-12. Questionnaires should take about 30 minutes total to complete.
  Other Names: Surveys
Device: Holter Monitor — Participants wear a Holter monitor for 20-24 hours to check nervous system and heart function at baseline and once during Days 3-7 and once during Days 8-12.
Other: Yogurt — Participants given 2 tablespoons (33 cc) of DannonÒ OikosÒ yogurt each day for 12 days.

SUMMARY:
The goal of this clinical research study is to learn if probiotics found in yogurt can help to decrease gastrointestinal (GI) symptoms in cancer patients. Probiotics are live bacteria and yeast that help with many of our functions and may help digestive problems. Researchers also want to learn if the bacteria in your stool change as your symptoms change while eating yogurt.

DETAILED DESCRIPTION:
Baseline Tests:

If you agree to take part in this study, you will have the following tests and procedures when you enroll:

* The coating on your tongue will be checked. Researchers think that the thickness of the coating on your tongue may be related to the microorganisms in your stomach and/or intestines.
* A stool sample will be collected for bacteria testing.
* You will be asked about your diet and how often you eat yogurt.
* You will wear a monitoring device called a Holter monitor for 20-24 hours to check your nervous system and heart function.
* You will be asked to complete 4 questionnaires about your symptoms in the past 24 hours, your irritable bowel syndrome (IBS), your most recent stool, and your quality-of-life. These questionnaires should take about 30 minutes total to complete.

Study Procedures:

One (1) time during Days 3-7 and 1 time during Days 8-12:

* You will be asked to complete the same 4 questionnaires you completed at baseline.
* A stool sample will be collected by your bedside nurse for bacteria testing.
* You may wear a Holter monitor to check your heart function.

You will be given at least 2 tablespoons (33 cc) of DannonÒ OikosÒyogurt each day.

Length of Study:

Your participation in this study will be over after you complete the study procedures during Days 8 to 12.

If you are discharged before you complete the study procedures above, you will be called and asked about your symptoms and given a stool collection kit. This phone call should take about 30 minutes to complete. The study staff will give you more information about stool collection. Your sample will be collected for bacteria testing at your next clinic visit.

This is an investigational study. The use of probiotics in yogurt to treat GI symptoms in cancer patients is investigational. The study doctor can explain how the probiotics are designed to work.

Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patient
2. 18 years old or older
3. Has gastrointestinal symptoms with severity score of </= 60 out of 100 visual analog scale for irritable bowel syndrome (VAS-IBS) in at least 2 out of 7 items measured
4. Able to eat by mouth
5. Estimated length of hospital stay is 10 days or more
6. Must give written study consent

Exclusion Criteria:

1. Neutropenic patient with absolute neutrophil count (ANC) less than 1000 cells/mm3
2. Patient within 100 days of auto /allo stem cell transplant and their stem cell physician does not approve yogurt ingestion.
3. Has intestinal obstruction.
4. Patient is currently on antibiotics
5. Allergic to yogurt
6. Patient who eats yogurt equal or more than once a day in the last 3 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Percentage Change in Bacteroidetes in Stool from Baseline to Day 12 | Baseline to Day 12
Percentage Change in Firmicutes in Stool from Baseline to Day 12 | Baseline to Day 12

SECONDARY OUTCOMES:
Adherence Rate of Dannon® Oikos® Yogurt Intake | 12 days
  Adherence rate calculated as percentage of times that a participant takes at least 2 table spoon (30 cc) of yogurt/day consumed for the 10±2 day prescription, as well as for the first 5±2 days, and will be summarized for each group using descriptive statistics. Regimen considered feasible for each group if at least 70% of participants in that group have reached at least 70% adherence rate in 10±2 days.

CONTACTS AND LOCATIONS:
Overall Officials: An T. Ngo-Huang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org